CLINICAL TRIAL: NCT03514264
Title: Clinical Applicability of PBSCIMMO as a Single Material in Endodontic Obturations
Acronym: PBSCIMMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Rubia Moura Leite Boczar, Principal investigator, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBS
Record Dates: First submitted 2018-02-26; First posted 2018-05-02 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Root Canal Therapy
Keywords: Endodontics; Biomaterials; Dental pulp cavity; Periapical abscess; Root canal therapy; Root canal obturation
MeSH Terms: conditions — Dental Caries; Periapical Abscess | interventions — Gutta-Percha

STUDY DESIGN:
Intervention Model Description: A randomized, interventional, prospective, unicentric, double blind clinical trial.
Who Masked: Outcomes Assessor
Masking Description: After 6 months the results will be evaluated by two independent professionals, who did not participate in the interventions and are not aware of the allocation. The evaluation will be performed by means of tomography and clinical examination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GUTTA PERCHA and AHPLUS cement (group A) (Experimental): 43 patients will undergo endodontic treatment with obturation with AHPlus cement and Gutta-Percha cones. This treatment will be performed in 2 sessions. First intervention: endodontic instrumentation and introduction of intra-canal medication that will remain in the tooth for 4 weeks. Second intervention: removal of intracanal medication and filling with cement and gutta percha AHPlus.
  Interventions: Procedure: Gutta Percha and AHPLUS cement (group A)
- PBS CIMMO cement (group B) (Experimental): 43 patients will undergo endodontic treatment with PBS CIMMO® cement (single material).This treatment will be performed in 1 session.Single intervention: endodontic instrumentation and cement filling PBS CIMMO.
  Interventions: Procedure: PBS CIMMO cement (group B)

INTERVENTIONS:
Procedure: Gutta Percha and AHPLUS cement (group A) — First intervention: endodontic instrumentation and introduction of intact medication that will remain inside the tooth for 4 weeks.
  Second intervention: removal of intracanal medication and canal filling with cement AHPLUS and guttapercha
  Arms: GUTTA PERCHA and AHPLUS cement (group A)
Procedure: PBS CIMMO cement (group B) — Single intervention: endodontic instrumentation and obturation with cement PBS CIMMO
  Arms: PBS CIMMO cement (group B)

SUMMARY:
A randomized, interventional, prospective, unicentric clinical study, 86 patients will be submitted to endodontic treatment of necrotic teeth. 43 patients will complete treatment with obturation with AHPlus cement and Gutta-Percha cones (group A) and 43 patients will complete treatment with PBS® CIMMO cement (single material) (group B). The primary outcome will be the repair of the periradicular lesion demonstrated by integrity of the hard blade throughout the perimeter of the root identified by Tomography Cone Beam, performed after 6 months of treatment. The secondary endpoint will be the absence of fistula after 6 months of treatment identified by clinical examination.

DETAILED DESCRIPTION:
GOALS PRIMARY OBJECTIVE-Evaluate the PBS CIMMO cement as a single element in endodontic obturations of necrotic teeth, through the analysis of integrity of the hard blade throughout the perimeter of the root of the treated tooth, identified by Tomography Cone Beam, after 6 months of treatment.

SECONDARY OBJECTIVE- Clinical evaluation of teeth treated after 6 months, with the purpose of identifying the absence of clinical signs and symptoms, through the finding of absence of fistula.

METHOD-DESIGN A randomized, interventional, prospective, unicentric, double blind clinical trial.

APPROVAL This work was approved by the Research Ethics Committee of the Vale do Sapucaí University (UNIVÁS) and is registered in the Brazilian Platform - Certificate of Approval for CAAE-number 77495717.7.0000.5102 CONSENT Relevant information from this study will be provided to all patients in an understandable way. Patients will have the opportunity to have their questions answered and will provide their consent by signing the free and informed consent form The study is being carried out in Brazil, in the urban area of the city of Pouso Alegre, state of Minas Geraes, in the Clinic of the Brazilian Association of Dentistry (ABO).

Interventions

The recommended techniques will be different for each group. GROUP A - CUTTING WITH CEMENT AHPLUS AND GUTTA HANGER

1. First session

   Intra-channel medication and instrumentation procedures:

   Local anesthesia with lidocaine and phenylephrine 1: 100,000 (DFL® Industry and Commerce-Brazil) will be used a tube containing 1.8 ml. Absolute insulation with clamp W8A and 8ª (SSWhite ® -Duflex-Brasil), rubber sheet (Madeitex®-Brazil) and arch (JON® Brazil). The opening will be performed with a high-speed motor (Dabi Atlante® Equipamentos Odontológicos Brasil), low rotation (Dabi Atlante®) and endodontic probe (Duflex®) drill 1016 HL (KG®-Sorensen). Mechanized instrumentation will be carried out using the Endo Easy SI® motor in reciprocating module. The endodontic instrument for instrumentation will be the Logic Easy® file numbering (2505). Pre-crown-down instrumentation will be performed on the cervical, middle and apical thirds, with apparent measurements determined by the initial radiograph. Each channel will receive irrigation with 2.5% sodium hypochlorite through a 10ml disposable syringe with a 0.55x20 24G hypodermic needle. 3/4 SR®. Then, the localization of the foramen with Novapex® foramen locator will be performed and the working length will be determined and then instrumentation with the same file will be determined. Through a reciprocating Easy Clean® device, PUI (Passive Ultrasonic Irrigation) with ethylene diamino tetraacetic acid, surfactant (EDTA T) Formula & Action® as well as sodium hypochlorite will be performed. Then, it will be installed in the channels, Callen PMCC SSWhite® (Calcium hydroxide paste with camphorated paramonoclorophenol) MIC (intra-canal medication) to perform disinfection of dentinal canaliculi. Such paste will temporarily seal these channels for 4 weeks.
2. Second session -After 30 days The obturation with AHPlus cement and Gutta Percha (group A) will be performed in 43 teeth, according to the following sequence: test of the main gutta percha Dentsply®, after foramen calibration. Handling of the AH Plus Dentsply® cement will be carried out. The medium cone will be greased with cement and taken to the canal. Through an Easy-Compressor term, the cone will be cut and compacted "hot" in the channel. New cone will be placed in the space conquered by compaction, will be cut "hot" by term compactor and then condensed by condenser instrument Schilder Oddus De Deus®. Soon after, the teeth will be restored with Charisma Kulzer® photopolymerizable resin, Radi® light curing. Patients will be submitted to final radiographs and receive systemic medication with analgesic Lisador® 1 tablet every 6 hours while there is pain. The recommended anti-inflammatory will be Decadron 4mg, 1 tablet every 12 hours for 3 days, if the patient can not use it, Maxulid 400 mg, 1 tablet every 12 hours for 3 days will be given. The antibiotic of choice will be Sinot Clav® 875 mg, 1 tablet every 12 hours for 7 days. In case of allergy to Amoxicillin, Dalacin 300 mg, 1 capsule every 8 hours for 7 days will be given. After 6 months, the patients will return to the Clinic of the Brazilian Association of Dentistry to perform a Cone Beam CT scan and clinical examination.

GROUP B - CUTTING WITH PBSCIMMO CEMENT SINGLE SESSION Instrumentation and filling procedures Local anesthesia with lidocaine and phenylephrine 1: 100,000 (DFL® Industry and Commerce-Brazil) will be used a tube containing 1.8 ml. Absolute insulation with clamp W8A and 8ª (SSWhite ® -Duflex-Brasil), rubber sheet (Madeitex®-Brazil) and arch (JON® Brazil). The opening will be performed with a high-speed motor (Dabi Atlante® Equipamentos Odontológicos Brasil), low rotation (Dabi Atlante®) and endodontic probe (Duflex®) drill 1016 HL (KG®-Sorensen). Mechanized instrumentation will be carried out using the Endo Easy SI® motor in reciprocating module. The endodontic instrument for instrumentation will be the Logic Easy® file numbering (2505). Pre-crown-down instrumentation will be performed on the cervical, middle and apical thirds, with apparent, determined by the initial radiography. Each channel will receive irrigation with 2.5% sodium hypochlorite through a 10ml disposable syringe with a 0.55x20 24G hypodermic needle. 3/4 SR®. Then, the localization of the foramen with Novapex® foramen locator will be performed and the working length will be determined and then instrumentation with the same file will be determined. Through a reciprocating Easy Clean® device, PUI (Passive Ultrasonic Irrigation) with ethylene diamino tetraacetic acid, surfactant (EDTA T) Formula & Action® as well as sodium hypochlorite will be performed. Continuously, the PBS CIMMO® cement will be installed in the channels, as a single obturator element. The CBS® PBS Cement seal (Group B) will be made of 43 teeth as follows: the instruments used will be the number 40 nickel and titanium Macspaden Flex Pack® micro-motor capacitors coupled to the internal dental office system and nickel and titanium in numbers and standard colors: Green (0.35 and 0.70), Black (0.40 and 0.80), Yellow (0.50 and 1.00), Blue (0.60 and 1.20). Handling of CIMMO® PBS cement will follow manufacturer's recommendations: on sterile glass plate, a portion of the cement powder and a drop of distilled water will be dispensed. Through a flexible spatula, the powder will be mixed to the liquid and spatulate until the consistency of toothpaste. The Macspaden Flex Pack® 40 instrument will then be coupled to the micro-motor and embedded in cement. When it is taken to the channel, the micro-motor will be activated and the channel will be in and out. Then, condensation will occur with the green condenser tip thinner and then thicker. In the same way, more cement will be brought to the channel with Flex Pack® number 40 and again condensed now with the black, thin point and then thick capacitors. These maneuvers will be repeated until the fine and thick blue capacitors are used and the absence of spaces is verified. Soon after, the teeth will be restored with Charisma Kulzer® photopolymerizable resin, Radi® light curing. Patients will be submitted to final radiographs and receive systemic medication with analgesic Lisador® 1 tablet every 6 hours while there is pain. The recommended anti-inflammatory will be Decadron®, 4mg, 1 tablet every 12 hours for 3 days, if the patient is unable to use it, Maxulid® 400mg, 1 tablet every 12 hours for 3 days will be given. The antibiotic of choice will be Sinot Clav® 875 mg, 1 tablet every 12 hours for 7 days. In case of allergy to Amoxicillin, Dalacin 300 mg, 1 capsule every 8 hours for 7 days will be given. After 6 months, the patients will return to the Clinic of the Associação Brasileira de Odontologia to perform a Cone Beam tomografy scan and clinical examination.

Sample size: 86 patients The observed response will be dichotomous, the type of analysis will be by comparing two proportions. The investigators accessed the site www.lee.dante.br 25, Lee-Samples for verification of possible identification of n. The proportions were based on the literature.

Proportion in group 1: 36% Proportion in group 2: 10% Level of significance: 5% Power of the test: 90% Hypothesis test: monocaudal Sample size calculated for each group: 43

Allocation: Patients are allocated to the study or control group in a 1: 1 ratio using a software-generated randomizer - RANDOMIZATION.COM (http://www.randomization.com)26. Concealment Mechanism: Opaque, sealed and serial number envelopes containing the group as well as the material to be used will be used to maintain the confidentiality of the random allocation. The envelopes will be delivered to the professional who performed the intervention at the initial moment Patients will not know which research group will participate. After 6 months, a CT scan and clinical examination will be performed. The evaluations will be performed by professionals who did not participate in the intervention and have more than 20 years of experience in endodontics. These professionals will not know to which group the patient belongs.

Recruitment of patients-waiting list of patients who seek the clinic of the Associação Brasileira de Odontologia (ABO) -UNIVÁS.

Beginning of appointments: November 2017 Data collection: June 2018.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with a diagnosis of necrosis.

Exclusion Criteria:

* Patients who drop out during the study
* Patients who do not return to the final exam after 6 months.
* Patients who present more than one tooth in need of treatment will choose only one tooth, the others will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-06-05 (Estimated); Study Completion 2019-02-26 (Estimated)

PRIMARY OUTCOMES:
Patients with necrotic teeth and periradicular lesion evaluated by cone beam tomography | Patients will return six months after the procedure to undergo a exam cone Beam tomografy
  The data will be aggregated by presence of hard blade that determines the phylogenetic parameter of success of the treatment. This physiological parameter is the presence of hard blade integrated in the tomography image, which will determine healthy periodontal ligament

SECONDARY OUTCOMES:
Clinical examination of patients' treated teeth | Patients will return six months after the procedure to undergo a clinical examination
  The physiological parameter for this examination will be the absence of fistula that will determine treatment success

CONTACTS AND LOCATIONS:
Overall Officials: Rubia Boczar, Principal Investigator — Univás-Universidade do Vale do Sapucaí- Pouso Alegre Minas Geraes; Taylor b Schnaider, MD,PhD, Study Director — Universidade Vale do Sapucaí; Daniela F Veiga, MD,PhD, Study Chair — Universidade Vale do Sapucaí
Locations (1):
- Rubia Moura Leite Boczar, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No